CLINICAL TRIAL: NCT06421740
Title: REal-world Utilization and Treatment Target ACHievement With Upadacitinib in Adolescents and Adults With Moderate to Severe Atopic Dermatitis in China
Brief Title: An Observational Study to Assess Real-World Use of Upadacitinib Tablets in Adolescent and Adult Participants With Moderate to Severe Atopic Dermatitis in China
Acronym: REACH-AD
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-965
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
Keywords: Upadacitinib; Rinvoq
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib: Participants will receive upadacitinib as prescribed by their physician according to local label.

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin.

Upadacitinib is an approved drug for treating AD. Approximately 1000 adolescents and adult participants who are prescribed upadacitinib by their physician in accordance with local label will be enrolled in up to 40 sites in China.

Participants will receive oral upadacitinib tablets as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed up for approximately 12 months.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (body weight >= 40 kg at the Baseline Visit for patients between >= 12 and < 18 years of age) and adults at the time of enrollment.
* Clinical diagnosis of moderate to severe atopic dermatitis at the time of enrollment.
* UPA treatment is indicated for AD and prescribed as per Chinese label / SmPC.
* The decision to prescribe UPA is made prior to and independent of study participation.
* The participant should not be treated with UPA prior to this study.
* Participants who are willing and able to participate in the collection of patient-reported data, including ePROs and eDiary via apps.
* The participant (legal representative for adolescents) voluntarily signed an informed consent before any study-related activities are conducted.

Exclusion Criteria:

* The participant is currently participating in interventional research (not including noninterventional study, observational study, or registry participation).
* Any circumstances that the investigator believes may limit the patient's participation and compliance with study procedures.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent and adult Chinese participants with atopic dermatitis (AD) who are prescribed Upadacitinib by their physician according to their local label.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a dose change | 12 Months
  Dose change includes: Changed dose, dose escalation or dose tapering.
Number of participants with interruption or permanent discontinuation | 12 Months
  Interruption: Upadacitinib is temporarily interrupted due to atopic dermatitis disease condition, economic, tolerance, AE, or personal reasons, and the investigator considers there is still possibility of Upadacitinib re-initiating within the patient's study follow-up period.
  Discontinuation: Upadacitinib is permanently discontinued for safety or any other reasons, and the investigator considers Upadacitinib will not be used again, at least within the participant's study follow-up period.
Number of participants with Upadacitinib drug compliance | 12 Months
  The participants missed medication, regardless of reason, or incompliance with the prescription as per medical advice are to be recorded in the eDiary, choosing the reason: "Forgot, Self-reduction of medication, interruption because of AE, interruption not due to safety/tolerability, for other reasons".
  If no eDiary entries are found within 30 days before the visit, the participant will need to complete the following question in ePRO: timely Upadacitinib intake per medical advice in past 30 days (yes/no); if "no", days-off-drug, intentionally or accidentally, and if "intentionally", reason for incompliance with medical prescription.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (38):
- China (38):
  - Beijing Anzhen Hospital /ID# 273443, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital /ID# 274778, Beijing, Beijing Municipality
  - Peking University First Hospital /ID# 274865, Beijing, Beijing Municipality
  - Peking Unversity Third hospital /ID# 274864, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital (East) - Dongdan Campus /ID# 264193, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Fujian Medical University /ID# 268210, Fuzhou, Fujian
  - Changgeng Hospital /ID# 268209, Xiamen, Fujian
  - Guangzhou Dermatology Hospital /ID# 271684, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital Of Sun Yat-Sen University /ID# 268618, Zhuhai, Guangdong
  - Hainan Fifth People's Hospital /ID# 269747, Hainan, Hainan
  - Hebei Engineering University Affiliated Hospital /ID# 268660, Handan, Hebei
  - The Second Affiliated Hospital Of Harbin Medical University /ID# 270872, Harbin, Heilongjiang
  - People's Hospital of Henan Province /ID# 269744, Zhengzhou, Henan
  - Wuhan Integrated TCM & Western Medicine Hospital（Wuhan No.1 Hospital) /ID# 272374, Wuhan, Hubei
  - Tongji Hospital /ID# 269745, Wuhan, Hubei
  - Xiangya Hospital Central South University /ID# 272373, Changsha, Hunan
  - Nanjing Drum Tower Hospital /ID# 268616, Nanjing, Jiangsu
  - Affiliated Hospital Of Nantong University /ID# 269743, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University /ID# 269742, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College /ID# 268208, Xuzhou, Jiangsu
  - Dalian Dermatosis Hospital /ID# 272495, Dalian, Liaoning
  - The People's Hospital of Liaoning Province /ID# 268206, Shenyang, Liaoning
  - Shandong Provincial Hospital /ID# 268661, Jinan, Shandong
  - Jining Medical University - Affiliated Hospital /ID# 270873, Jining, Shandong
  - Weifang People'S Hospital /ID# 268659, Weifang, Shandong
  - Ruijin Hospital /ID# 268658, Shanghai, Shanghai Municipality
  - Huashan Hospital Of Fudan University /ID# 270277, Shanghai, Shanghai Municipality
  - Shanghai Sixth People'S Hospital /ID# 268617, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital /ID# 268657, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University /ID# 268313, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital /ID# 268314, Chengdu, Sichuan
  - The Affiliated Hospital Of Southwest Medical University /ID# 268207, Sichuan, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region /ID# 269746, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical College /ID# 273451, Kunming, Yunnan
  - Zhejiang Provincial Hospital of Chinese Medicine /ID# 268613, Hangzhou, Zhejiang
  - Ningbo No.6 hospital /ID# 268315, Ningbo, Zhejiang
  - Taizhou Central Hospital /ID# 268211, Taizhou, Zhejiang
  - Zhuji People'S Hospital /ID# 268614, Zhuji, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-965